CLINICAL TRIAL: NCT01145196
Title: Genotype - Phenotype Study of Patients With Plaquenil-induced Retinal Toxicity
Brief Title: Genotype-Phenotype Study of Patients With Plaquenil -Induced Retinal Toxicity, With Evaluation of the ABCA4 Gene
Status: Recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100140; 10-EI-0140
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-10-24

CONDITIONS: Genotype; Retinal Disease
Keywords: Retinal Disease; Plaquenil-Induced; Natural History
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected: Participants affected by Plaquenil induced retinal toxicity
- Unaffected: control participants without Plaquenil induced retinal toxicity

SUMMARY:
Background:

- Plaquenil (hydroxychloroquine) is an anti-inflammatory drug that is used to treat some autoimmune diseases such as lupus and rheumatoid arthritis. This drug can damage the retina by causing a condition called plaquenil-induced retinal toxicity, which may lead to vision loss. However, most people taking plaquenil do not develop this problem. Researchers are interested in studying whether differences in a person s genes explain why some people develop plaquenil-induced retinal toxicity while others do not.

Objectives:

- To investigate possible correlations between certain genes or genetic mutations and plaquenil-induced retinal toxicity.

Eligibility:

* Individuals at least 18 years of age who have previously used plaquenil.
* Both individuals who have and have not developed plaquenil-induced retinal toxicity will be eligible for this study.

Design:

* The study requires one or two visits to the National Eye Institute or an outpatient study clinic over a maximum 2-year period.
* Participants will provide a personal and family medical history, and will have a full eye examination.
* Participants will also provide blood samples for testing.
* No treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
OBJECTIVE:

The objective of this study is to investigate whether there is a correlation between genetic mutations, beginning with an analysis of ABCA4, and Plaquenil(R)-induced retinal toxicity and to describe the phenotype of Plaquenil(R)-induced retinal toxicity.

STUDY POPULATION:

The study will enroll 100 patients, 18 years of age or older, found to have Plaquenil(R)-induced retinal toxicity. 200 volunteers with systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), or Sj(SqrRoot)(Delta)gren s syndrome and history of Plaquenil(R) use, but without evidence of retinal toxicity, will also be recruited.

DESIGN:

The study is an observational study with 1-2 outpatient visits to the NEI clinic or review of medical records for off-site participants. All participants will provide a blood sample for genetic analysis.

OUTCOME MEASURES:

Clinical examination and blood samples will be used for genetic testing and mutation identification. The primary outcome of this study is to identify genetic mutations, starting with those in ABCA4 gene, associated with retinal toxicity in participants with a history of Plaquenil(R) use. Secondary objectives include determining the utility of testing metrics in evaluating the presence of retinal toxicity.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Affected participants must be 18 years of age or older and have:

   * History of systemic lupus erythematosus (SLE), rheumatoid arthritis (RA) or Sj(SqrRoot)(Delta)gren s syndrome, and
   * History of Plaquenil use, and
   * Evidence of Plaquenil -induced retinal toxicity, based on clinical findings.
2. Unaffected volunteers must be 18 years of age or older and have:

   * History of systemic lupus erythematosus (SLE), rheumatoid arthritis (RA) or Sj(SqrRoot)(Delta)gren s syndrome, and
   * History of Plaquenil use, and
   * No retinal disease upon examination within the last six months.
3. All participants must be able to:

   * Provide their own consent, and
   * Safely provide a blood sample.

<TAB>

EXCLUSION CRITERIA:

1. Participants with other known (genetic) retinal disease including but not limited to: Stargardt s disease and cone or cone-rod dystrophy whose diagnosis preceded their Plaquenil use. Participants with no known previous genetic diagnosis but with clinical findings associated with a genetic diagnosis, such as parafoveal or macular flecks which are associated with Stargardt s disease or fundus flavimaculatus, will also be excluded.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll 100 patients, 18 years of age or older, found to have Plaquenil -induced retinal toxicity. 200 volunteers with systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), or Sjogren's syndrome and history of Plaquenil use, but without evidence of retinal toxicity, will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2010-08-23 (Actual)

PRIMARY OUTCOMES:
The outcome of this study is to identify genetic mutations, starting with those in ABCA4 gene, associated with retinal toxicity in participants with a history of plaquenil use. | annually for five years
  The outcome of this study is to identify genetic mutations, starting with those in ABCA4 gene, associated with retinal toxicity in participants with a history of plaquenil use.

SECONDARY OUTCOMES:
The secondary outcome of this study is to determine the utility of various testing metrics in evaluating the presence of retinal toxicity. | annually for five years
  The secondary outcome of this study is to determine the utility of various testing metrics in evaluating the presence of retinal toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy GD, Munz SJ, Paschal J, Cohen HB, Pince KJ, Peterson T. Incidence of hydroxychloroquine retinopathy in 1,207 patients in a large multicenter outpatient practice. Arthritis Rheum. 1997 Aug;40(8):1482-6. doi: 10.1002/art.1780400817. PMID 9259429
- [Background] HOBBS HE, SORSBY A, FREEDMAN A. Retinopathy following chloroquine therapy. Lancet. 1959 Oct 3;2(7101):478-80. doi: 10.1016/s0140-6736(59)90604-x. No abstract available. PMID 14402143
- [Background] Webster AR, Heon E, Lotery AJ, Vandenburgh K, Casavant TL, Oh KT, Beck G, Fishman GA, Lam BL, Levin A, Heckenlively JR, Jacobson SG, Weleber RG, Sheffield VC, Stone EM. An analysis of allelic variation in the ABCA4 gene. Invest Ophthalmol Vis Sci. 2001 May;42(6):1179-89. PMID 11328725
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-EI-0140.html